CLINICAL TRIAL: NCT05304780
Title: Effectiveness of a Needs-tailored Nurse-led Recovery Program for Community-dwelling People With Schizophrenia: A Cluster-randomized Controlled Trial
Brief Title: Needs-tailored Nurse-led Recovery Program for Community-dwelling People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wen I Liu, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: needs-tailored
Record Dates: First submitted 2022-03-03; First posted 2022-03-31 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Schizophrenia; Recovery; Medication Adherence
Keywords: Needs-tailored; Recovery; Empowerment; Hope; Medication Adherence; Cluster-randomized controlled trial
MeSH Terms: conditions — Schizophrenia; Medication Adherence; Empowerment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Needs-tailored nurse-led recovery program
  Interventions: Behavioral: needs-tailored nurse-led recovery program
- Control group (No Intervention): existing community homecare services

INTERVENTIONS:
Behavioral: needs-tailored nurse-led recovery program — The needs-tailored nurse-led recovery program were divided into five major stages of care, which were build partnership, conduct integrated needs assessment, set needs-based recovery goals and provide empowerment-oriented care, conduct continuous monitoring of goals, and conduct effectiveness evaluations.
  Arms: experimental group

SUMMARY:
Meeting people's needs is positively correlated with their recovery. However, recovery services rarely include nurse-led programs tailored to the needs of these people. This study aimed to evaluate the effectiveness of a new needs-tailored recovery program by using a cluster-randomized controlled trial design.

DETAILED DESCRIPTION:
First year, investigators used the pilot study to test the needs tailored recovery program feasibility, acceptability and preliminary usefulness of the needs-tailored nurse-led recovery program. In the second year, based on the findings of the pilot study, a cluster randomized controlled trial was conducted to assess the effectiveness of the needs-tailored nurse-led recovery program in two psychiatric centers in northern Taiwan. The treatment group receive the needs-tailored nurse-led recovery program by their home-care nurses over 6 months. The control group receive the usual community psychiatric care only. Data were collected before the intervention, after the intervention, and at a follow-up session three months after the end of the intervention period. The outcomes were recovery, needs, hope, empowerment, psychotic symptoms, and medication adherence. The investigators used repeated measures ANOVA tests to examine the effect of the group × time interaction.

ELIGIBILITY:
Inclusion Criteria:

* were living in the community and had a diagnosis of schizophrenia based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* were aged 20-64 years
* were able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* were living in a community institution such as a recovery home, community rehabilitation center, nursing home, or day hospital
* had a neurocognitive disorder, substance abuse disorder, or comorbidity.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change scores of Questionnaire about the Process of Recovery | baseline
  Participants will complete the Questionnaire about the Process of Recovery (QPR). It is total of 22 questions in this scale to evaluate recovery score.Each question is scored from 0-4 points.The higher scores mean a better outcome.
Change scores of Questionnaire about the Process of Recovery | 6 months
  Participants will complete the Questionnaire about the Process of Recovery (QPR). It is total of 22 questions in this scale to evaluate recovery score.Each question is scored from 0-4 points.The higher scores mean a better outcome.
Change scores of Questionnaire about the Process of Recovery | 9 months
  Participants will complete the Questionnaire about the Process of Recovery (QPR). It is total of 22 questions in this scale to evaluate recovery score.Each question is scored from 0-4 points.The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change scores of Rogers Empowerment Scale | baseline
  Participants will complete the Empowerment Scale. It is total of 13 questions in this scale to evaluate empowerment score. Each question is scored from 1-4 points.The higher scores mean a better outcome.
Change scores of Rogers Empowerment Scale | 6 months
  Participants will complete the Empowerment Scale. It is total of 13 questions in this scale to evaluate empowerment score. Each question is scored from 1-4 points.The higher scores mean a better outcome.
Change scores of Rogers Empowerment Scale | 9 months
  Participants will complete the Empowerment Scale. It is total of 13 questions in this scale to evaluate empowerment score. Each question is scored from 1-4 points.The higher scores mean a better outcome.
Change scores of Needs Assessment Instrument for the Community-Dwelling People with Mental Illness | baseline
  Participants will complete the Needs Assessment Instrument for the Community-Dwelling People with Mental Illness. It is total of 22 questions in this scale to evaluate need. Each question is scored from 0-2 points. The higher the score, the greater the demand.
Change scores of Needs Assessment Instrument for the Community-Dwelling People with Mental Illness | 6 months
  Participants will complete the Needs Assessment Instrument for the Community-Dwelling People with Mental Illness. It is total of 22 questions in this scale to evaluate need. Each question is scored from 0-2 points. The higher the score, the greater the demand.
Change scores of Needs Assessment Instrument for the Community-Dwelling People with Mental Illness | 9 months
  Participants will complete the Needs Assessment Instrument for the Community-Dwelling People with Mental Illness. It is total of 22 questions in this scale to evaluate need. Each question is scored from 0-2 points. The higher the score, the greater the demand.
Change scores of Herth Hope Index | baseline
  Participants will complete the Herth Hope Index (HHI). It is total of 12 questions in this scale to evaluate hope score.Each question is scored from 1-4 points.The higher scores mean a better outcome.
Change scores of Herth Hope Index | 6 months
  Participants will complete the Herth Hope Index (HHI). It is total of 12 questions in this scale to evaluate hope score.Each question is scored from 1-4 points.The higher scores mean a better outcome.
Change scores of Herth Hope Index | 9 months
  Participants will complete the Herth Hope Index (HHI). It is total of 12 questions in this scale to evaluate hope score.Each question is scored from 1-4 points.The higher scores mean a better outcome.
Change scores of Medication Adherence Rating Scale | baseline
  Participants will complete the Medication Adherence Rating Scale (MARS). It is total of 10 questions in this scale to evaluate medication adherence score. Each question is scored from 0-1 points.The higher scores mean a better outcome.
Change scores of Medication Adherence Rating Scale | 6 months
  Participants will complete the Medication Adherence Rating Scale (MARS). It is total of 10 questions in this scale to evaluate medication adherence score. Each question is scored from 0-1 points.The higher scores mean a better outcome.
Change scores of Medication Adherence Rating Scale | 9 months
  Participants will complete the Medication Adherence Rating Scale (MARS). It is total of 10 questions in this scale to evaluate medication adherence score. Each question is scored from 0-1 points.The higher scores mean a better outcome.
Change scores of Brief Psychiatric Rating Scale | baseline
  Participants will complete the Brief Psychiatric Rating Scale (BPRS). It is total of 16 questions in this scale to evaluate psychiatric symptom. Each question is scored from 0-6 points.The higher scores mean a worse outcome.
Change scores of Brief Psychiatric Rating Scale | 6 months
  Participants will complete the Brief Psychiatric Rating Scale (BPRS). It is total of 16 questions in this scale to evaluate psychiatric symptom. Each question is scored from 0-6 points.The higher scores mean a worse outcome.
Change scores of Brief Psychiatric Rating Scale | 9 months
  Participants will complete the Brief Psychiatric Rating Scale (BPRS). It is total of 16 questions in this scale to evaluate psychiatric symptom. Each question is scored from 0-6 points.The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu WI, Hsieh WL, Lai CT, Liu CC, Tai YM, Liu CY. Effectiveness of a needs-tailored nurse-led recovery program for community-dwelling people with schizophrenia: a cluster-randomized controlled trial. BMC Nurs. 2024 May 16;23(1):329. doi: 10.1186/s12912-024-01986-x. PMID 38755582